CLINICAL TRIAL: NCT05576129
Title: Theta-gamma Transcranial Alternating Current Stimulation (tACS) to Modulate Activity in Sensorimotor Cortex for Improvement of Motor Skill Acquisition in Stroke Patients
Brief Title: Transcranial Alternating Current Stimulation (tACS) to Improve Motor Skill Acquisition in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Technical University of Twente (Other); University of Oxford (Other)
Responsible Party: Principal Investigator, Fanny Quandt, Principal Investigator, Universitätsklinikum Hamburg-Eppendorf
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: CFC_tACS_Stroke
Record Dates: First submitted 2022-10-07; First posted 2022-10-12 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Stroke
Keywords: Stroke; Hand motor impairment; Transcranial alternating current stimulation; Non-invasive brain stimulation; motor learning; sensorimotor cortex; crossfrequency coupling; theta-gamma phase amplitude coupling
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TGP-tACS (Active Comparator): Patients perform a motor skill acquisition task with the affected hand during TGP-stimulation over the sensorimotor cortex on the lesioned side.
  Interventions: Device: TGP-tACS
- Sham-tACS (Sham Comparator): Patients perform a motor skill acquisition task with the affected hand during sham-stimulation over the sensorimotor cortex on the lesioned side.
  Interventions: Device: Sham-tACS

INTERVENTIONS:
Device: TGP-tACS — 38 min and 20s of 4mA peak-to-peak theta-gamma stimulation with 75 Hz-gamma coupled to the peak of 6Hz-theta waves. 3s ramp-up at the beginning of stimulation and 3s ramp-down at the end of stimulation.
  Administered using a Starstim® device and 5 gel electrodes with a πcm² area.
  Arms: TGP-tACS
Device: Sham-tACS — 38 min and 20s of alternation between 10s of 4mA peak-to-peak TGP- tACS and a 6 min 30s stimulation-free interval. Each stimulation consists of 3s ramp-up, 4s TGP stimulation and 3s ramp-down. Administered using a Starstim® device and 5 gel electrodes with a πcm² area.
  Arms: Sham-tACS

SUMMARY:
Hand motor function is often severely affected in stroke patients and its recovery is one primary goal in stroke rehabilitative treatment programs. Recently, theta-gamma transcranial alternating current stimulation (tACS) has been shown to enhance motor skill acquisition in healthy individuals. The aim of the present study is to examine the effect of theta-gamma tACS on motor skill acquisition in chronic stroke patients.

DETAILED DESCRIPTION:
Hand motor function is often severely affected in stroke patients and recovery of function is a primary goal in stroke rehabilitative treatment programs. Recently, theta-gamma tACS has been shown to enhance motor skill acquisition in healthy individuals [Akkad et al.2021]. The aim of the present study is to examine the effect of theta-gamma tACS on motor skill acquisition in chronic stroke patients.

In a randomized, controlled, triple-blind trial, chronic stroke patients with an initially impaired hand motor function will receive either (i) theta-gamma peak stimulation (TGP) or (ii) sham stimulation. TGP stimulation significantly improved motor learning in the study by Akkad et al (2021) compared to sham stimulation. tACS will be delivered through a five-electrode montage centered over the sensorimotor cortex on the lesioned side of the brain for approximately 38 min. During stimulation patients will perform a motor skill acquisition task performed with the affected hand. The task consists of short repetitive trials in which participants alternately press two buttons with their thumb. It is designed in a way that participants can improve their performance, more precisely the speed of button presses, and are encouraged to do so. To reduce skin sensations beneath the stimulation electrodes and thereby improve blinding compared to sham stimulation, a local anesthetic consisting of lidocaine and prilocaine will be administered underneath the stimulation electrodes.

Based on the results of the study by Akkad et al. (2021) and on the assumption that theta-gamma phase amplitude coupling is a key mechanism for motor skill acquisition, the investigators hypothesize that motor skill acquisition will differ significantly between the TGP and sham group.

ELIGIBILITY:
Inclusion Criteria:

* German-speaking
* ability to perform a thumb movement task with the affected hand
* first-ever clinical ischemic stroke in the chronic phase
* persistent mild motor deficit of the upper extremity or motor deficit of the upper extremity in the acute phase over >24h

Exclusion Criteria:

* pronounced cognitive deficits
* history of major neurological or psychiatric illness other than stroke
* epilepsy or epileptic seizure in the history
* any devices or implants in the head region (e.g. cochlear implant, aneurysm clips),
* implanted pacemaker or medical pumps
* intake of psychotropic medication
* allergy to any ingredient of the local anesthetic cream
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-11-14 (Actual); Primary Completion 2023-08-25 (Actual); Study Completion 2023-08-25 (Actual)

PRIMARY OUTCOMES:
Motor Skill Acquisition | Over the course of the motor task with a duration of 38 minutes and 20 seconds.
  Quotient of mean "Duration of Button Presses" of the best block and the baseline block. Best block is defined as the block with the lowest mean "Duration of Button Presses". "Duration of Button Press" is the Duration between the first and fourth button press of a valid trial.

SECONDARY OUTCOMES:
Duration of Button Presses | Baseline (consisting of 20 trials) and each of 6 blocks (consisting of 40 trials each)
  Time span from first to last button press of a trial. Averaged for all trials of one block

OTHER OUTCOMES:
"Thumb Speed" and "Thumb Acceleration" | Over the course of the motor task with a duration of 38 minutes and 20 seconds.
  An accelerometer will be fixed to the medial distal phalanx of the thumb. It measures the thumb acceleration in all three dimensions of space. We will use the accelerometer data for post-hoc explorative analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Fanny Quandt, Dr., Principal Investigator — Department of Neurology; University Medical Center Hamburg-Eppendorf; Bettina Schwab, PhD, Principal Investigator — Biomedical Signals and Systems, Technical Medical Centre, University of Twente, The Netherlands
Locations (1):
- Department of Neurology, University Medical Center Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared after main publication of results

REFERENCES:
- [Background] Akkad H, Dupont-Hadwen J, Kane E, Evans C, Barrett L, Frese A, Tetkovic I, Bestmann S, Stagg CJ. Increasing human motor skill acquisition by driving theta-gamma coupling. Elife. 2021 Nov 23;10:e67355. doi: 10.7554/eLife.67355. PMID 34812140
- [Result] Grigutsch LS, Haverland B, Timmsen LS, Asmussen L, Braass H, Wolf S, Luu TV, Stagg CJ, Schulz R, Quandt F, Schwab BC. Differential effects of theta-gamma tACS on motor skill acquisition in young individuals and stroke survivors: A double-blind, randomized, sham-controlled study. Brain Stimul. 2024 Sep-Oct;17(5):1076-1085. doi: 10.1016/j.brs.2024.09.001. Epub 2024 Sep 6. PMID 39245294